CLINICAL TRIAL: NCT00127829
Title: A Phase I, Open-Label, Dose Escalation Study Evaluating High-Dose Gefitinib (IRESSA®) on Weekly and Twice Weekly Schedules in Subjects With Solid Malignancies That Are Locally Advanced, Recurrent or Metastatic
Brief Title: Study Evaluating Gefitinib (IRESSA®) in Subjects With Solid Malignancies That Are Locally Advanced, Recurrent or Metastatic
Acronym: AGUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Alison Armour, MD, IRESSA Medical Science Director, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7913C00022
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Tumors
Keywords: Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Gefitinib

ARMS (1):
- 1 (Experimental): Gefitinib (IRESSA®)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Oral tablet
  Other Names: IRESSA®

SUMMARY:
This study will determine the safety profile and maximum tolerated dose (MTD) of orally administered gefitinib on a weekly and twice weekly schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor refractory to conventional treatment or whom no standard of treatment exists
* Life expectancy of > 12 weeks
* World Health Organization (WHO) performance status of < 2

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib or any of the excipients of this product
* Less than 4 weeks since completion of prior chemotherapy or radiation therapy (except nitrosoureas or mitomycin-C which must have a wash out period of 6 weeks)
* Incomplete healing from previous oncologic or other major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2005-07; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California